CLINICAL TRIAL: NCT00151827
Title: Efficacy and Safety of Olmesartan Medoxomil Compared With Losartan in Patients With Hypertension and Mild to Moderate Renal Impairment
Brief Title: Olmesartan Medoxomil in Hypertension and Renal Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sankyo Pharma Gmbh (Industry)
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SE-866/43
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Essential Hypertension; Renal Impairment
MeSH Terms: conditions — Essential Hypertension; Renal Insufficiency | interventions — Olmesartan Medoxomil; Losartan; Furosemide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olmesartan medoxomil (Experimental): Olmesartan oral tablets 20 mg or 40 mg + losartan placebo. Medications are taken once daily before breakfast with water.
  Interventions: Drug: Olmesartan medoxomil; Drug: Furosemide oral tablets
- Losartan (Experimental): Losartan over encapsulated tablets 50 mg and 100 mg plus olmesartan placebo.
  Interventions: Drug: Losartan; Drug: Furosemide oral tablets

INTERVENTIONS:
Drug: Olmesartan medoxomil — Olmesartan oral tablets 20 or 40 mg + losartan placebo. Medications are taken once daily before breakfast with water.
  Arms: Olmesartan medoxomil
Drug: Losartan — Medications are taken once daily before breakfast with water.
  Arms: Losartan
Drug: Furosemide oral tablets — If its use is necessary, the dose of furosemide allowed is 20 to 120 mg per day at the discretion of the investigator

SUMMARY:
This is a study in hypertensive patients with mild to moderate renal impairment. The antihypertensive efficacy of olmesartan medoxomil is compared to losartan.

ELIGIBILITY:
Inclusion Criteria:

* Mean sitting BP prior to randomization of 140-180/90-109 mmHg;
* Renal impairment prior to randomization of mild (50 ≤ CLcr ≥ 80 mL/min) to moderate (30 ≤ CLcr ≥50 mL/min) severity

Exclusion Criteria:

* Malignant hypertension or sitting BP greater than 180/109 mmHg;
* Severe heart failure, severe renal disease;
* Recent history of myocardial infarction, stroke or transient ischemic attack;
* History, clinical or current evidence of any significant gastrointestinal, respiratory, hematological, metabolic, immunological or any other underlying disease which in the opinion of the investigator would interfere with the patient's participation in the trial;
* Hypersensitivity or contraindications to ARBs or ACE inhibitors or any cross allergy;
* Treatment with dis-allowed medication;
* Pregnant or breastfeeding females or females of childbearing potential without adequate contraception;
* History of drug and/or alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2003-08; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Change in mean sitting diastolic blood pressure (dBP), assessed by conventional blood pressure measurements after 12 weeks of treatment | Baseline to 12 weeks

SECONDARY OUTCOMES:
Change in mean sitting diastolic blood pressure, assessed by conventional blood pressure measurements after 1, 2, 3, 8, 18, 24, 30, 36, 44 and 52 weeks of treatment; | Baseline to 1, 2, 3, 8, 18, 24, 30, 36, 44 and 52 weeks
Change in mean sitting systolic blood pressure, assessed by conventional blood pressure measurements after 1, 2, 3, 8, 18, 24, 30, 36, 44 and 52 weeks of treatment; | Baseline to 1, 2, 3, 8, 18, 24, 30, 36, 44 and 52 weeks
Response to treatment after 1, 2, 4, 8, 12, 18, 24, 30, 36, 44 and 52 weeks of treatment; | Baseline to 1, 2, 4, 8, 12, 18, 24, 30, 36, 44 and 52 weeks
  Response to treatment = mean sitting diastolic blood pressure less than or equal to 90 mmHg or reduction greater than or equal to 10 mmHg
Changes in creatinine clearance after 12 and 52 weeks of treatment, changes in proteinuria after 4, 12, 24, 36 and 52 weeks of treatment; | Baseline to 12 and 52 weeks
Changes in serum creatinine after 12 and 52 weeks of treatment | Baseline to 12 and 52 weeks
Rate of patients per dose level after 12 and 52 weeks of treatment | Baseline to 12 and 52 weeks
Change in proteinuria after 4, 12, 24, 36 and 52 weeks of treatment | Baseline to 4, 12, 24, 36 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: P. U. Witte, MD, PhD, Principal Investigator — IMFORM GmbH, Darmstadt, Germany
Locations (1):
- Darmstadt, Germany